CLINICAL TRIAL: NCT00284765
Title: Optimation of Treatment of the Sprained Ankle by Help of NSAID-Plaster (Flector). A Questionnaire.
Brief Title: Management of the Sprained Ankle by Help of NSAID-Plaster
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kolding Sygehus (Other)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: VF-20050182
Record Dates: First submitted 2006-01-31; First posted 2006-02-01 (Estimated); Last update posted 2006-03-13 (Estimated); Status verified 2006-01

CONDITIONS: The Sprained Ankle
MeSH Terms: interventions — diclofenac hydroxyethylpyrrolidine

INTERVENTIONS:
Procedure: flector

SUMMARY:
The purpose of this trial is to study the management of the sprained ankle by help of NSAID-plaster. A questionnaire. The effect of RICE and RICE + NSAID-plaster in the treatment of the sprained ankle, compared by pain-score.

ELIGIBILITY:
Inclusion Criteria:

* A sprained ankle, less than 24 hours old, understanding Danish, 18 years or older

Exclusion Criteria:

* Fracture of the ankle, wound around the ankle, allergy of NSAID- pregnancy, daily use of NSAID, GI-bleeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 2006-02; Study Completion 2006-05

PRIMARY OUTCOMES:
Pain-score

CONTACTS AND LOCATIONS:
Overall Officials: Berit Jørgensen, MD, Principal Investigator — Kolding Sygehus
Locations (1):
- Kolding Sygehus, Kolding, Denmark